CLINICAL TRIAL: NCT06898268
Title: Efficacy and Safety of Ondansetron Versus Metaclopromide Treatment in Infants With Gastro Oesophageal Reflux, a Comparative Study of Short Trial.
Brief Title: Efficacy and Safety of Ondansetron Versus Metaclopromide Treatment in Infants With Gastro Oesophageal Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRIRUMDGKHAN
Record Dates: First submitted 2025-03-22; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Reflux Disorder
MeSH Terms: interventions — Metoclopramide; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metoclopramide group (Experimental): Patients were prescribed metoclopramide twice a day for one week.
  Interventions: Drug: Metoclopramide
- Ondansetron (Experimental): Patients in this group were put on oral ondansetron in BD doses for one week.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Metoclopramide — Patients were prescribed metoclopramide twice a day for one week.
  Arms: Metoclopramide group
Drug: Ondansetron — Patients were put on oral ondansetron in BD doses for one week.
  Arms: Ondansetron

SUMMARY:
This study aimed to fill the gaps by comparing the efficacy and safety of ondansetron versus metoclopramide for the control of gastroesophageal reflux disorder in children 1-12 months of age, presenting at the outdoor department of Allama Iqbal Teaching Hospital, Dera Ghazi Khan.

DETAILED DESCRIPTION:
Since the FDA issued a warning against domperidone as a potential proarrhythmic drug in children, its use has been widely discouraged and no longer recommended in safe practices. This warning at one end persuaded the pediatricians to search for the new options; on the other end, the use of metoclopramide, H2 receptor antagonists, and alginate-based medications became superfluous, opening a wide area of research in search of the next potential best option. The findings of this study would add to the existing statistics and help clinicians to have better outcomes among infants with gastroesophageal reflux disorder.

ELIGIBILITY:
Inclusion Criteria:

* Infants of any gender
* Aged 1-12 months
* Presenting with symptoms of gastroesophageal reflux disease not responding to dietary modifications and positioning
* Afebrile at the time of presentation
* Vitally stable

Exclusion Criteria:

* No evidence of hypertrophic pyloric stenosis on ultrasonography
* Children with congenital heart disease
* Any history of prior illness associated with symptoms
* With abdominal distension
* Neurological impairment, like developmentally delayed, grossly microcephalic

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 1 week
  Reduction in vomiting episodes and preservation/increase in previous weight
Treatment-emerged adverse events | 1 week
  The occurrence of diarrhea, constipation, lethargy/somnolence, dark urine, headache, and warm flushes was considered as treatment-emerged adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Irum Jabeen, FCPS, Principal Investigator — Allama Iqbal Teaching Hospital, Dera Ghazi Khan, Pakistan; Asma Akbar, FCPS, Principal Investigator — Allama Iqbal Teaching Hospital, Dera Ghazi Khan, Pakistan
Locations (1):
- Allama Iqbal Teaching Hospital, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
If a reasonable request is made, data can be shared.